CLINICAL TRIAL: NCT04889534
Title: Evaluation of Predictive Factors for Nausea, Vomiting and Postoperative Acute Pain in Oncological Patients
Brief Title: Predictive Factors for Postoperative Pain, Nausea and Vomiting in Oncological Patients
Acronym: PONV
Status: Completed | Type: Observational
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Collaborators: Sponsor GmbH (Other)
Responsible Party: Sponsor
Other Study IDs: NP380/2013
Record Dates: First submitted 2018-08-09; First posted 2021-05-17 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2015-02

CONDITIONS: Nausea; Vomiting; Pain, Postoperative
Keywords: nausea; vomiting; pain
MeSH Terms: conditions — Nausea; Vomiting; Pain, Postoperative; Pain | interventions — Analgesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Analgesia — Patients will be observed during postoperative period,

SUMMARY:
1809 patients were evaluated in postoperative period. They were asked about nausea, vomiting, retching and pain in the first postoperative 24 hours

DETAILED DESCRIPTION:
Patients were prospectively evaluated , and nausea, vomiting and pain were recorded.

ELIGIBILITY:
Inclusion Criteria:

* patients submitted to oncological surgeries

Exclusion Criteria:

* refusal to sign the agreement term
* lack of information in the records

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients submitted to oncological surgeries in a specialized Hospital
Sampling Method: Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2015-01; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Intensity of postoperative pain | 24 hours
  pain intensity was measured using descriptive and verbal number scale

SECONDARY OUTCOMES:
side effects from analgesia | 24 hours
  nausea, vomiting, pruritus and hypotension were measured during first 24 postoperative hours

CONTACTS AND LOCATIONS:
Overall Officials: Hazem A Ashmawi, phD, Study Director — University of Sao Paulo
Locations (1):
- Angela Maria Sousa, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Lee SY, Hung CJ, Chen CC, Wu CC. Survival analysis of postoperative nausea and vomiting in patients receiving patient-controlled epidural analgesia. J Chin Med Assoc. 2014 Nov;77(11):589-93. doi: 10.1016/j.jcma.2014.08.008. Epub 2014 Sep 22. PMID 25249302
- [Background] Gramke HF, de Rijke JM, van Kleef M, Kessels AG, Peters ML, Sommer M, Marcus MA. Predictive factors of postoperative pain after day-case surgery. Clin J Pain. 2009 Jul-Aug;25(6):455-60. doi: 10.1097/AJP.0b013e31819a6e34. PMID 19542791